CLINICAL TRIAL: NCT02588703
Title: Delivering Treatment in DUI Programs to Reduce Alcohol-Related Disparities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Principal Investigator, Karen Osilla, Senior Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MD007762 (NIH)
Record Dates: First submitted 2015-08-17; First posted 2015-10-28 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): 9-session 2-hour group cognitive behavioral therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Usual Care (Active Comparator): 9-session 2-hour group counseling
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Coping Skills Treatment
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy
Behavioral: Usual Care — Existing DUI program group counseling
  Arms: Usual Care

SUMMARY:
The current study evaluates the efficacy of Cognitive Behavioral Therapy (CBT) in DUI programs for individuals with a first-time offense. Investigators will utilize a two-group randomized design where individuals enrolled in a DUI program with a first-time conviction will be randomized to Cognitive Behavioral Therapy (CBT; n=150) or Usual Care (UC; n=150). Participants will be assessed at baseline, immediately post-treatment, and 6-months post-treatment. Recidivism data will also be collected using administrative data two years post-treatment.

DETAILED DESCRIPTION:
Enormous unmet needs for alcohol treatment exist among individuals convicted of driving under the influence (DUI) since up to 43% recidivate and 67% meet criteria for alcohol dependence. Investigators will test whether delivering a cognitive behavioral treatment (CBT) for alcohol use disorders (AUDs) as part of a mandated DUI program improves health outcomes, and reduces alcohol use, alcohol-related problems and injuries, and DUI recidivism compared to usual care. The study has the potential to promote the public welfare by providing treatment to individuals with a DUI conviction, while focusing on Latinos, who are disproportionately less likely to access treatment and more likely to be arrested for a DUI, to have higher rates of recidivism, and to die in alcohol-related crashes than their white counterparts. The study is innovative because it would be the first to address effectiveness of treatment for AUDs embedded within a DUI program. Investigators will conduct a randomized trial of a 9-session group-based CBT (n=150) as compared to group-based usual care (UC; n=150) immediately after and 6 months after the end of treatment. Short-term outcomes include alcohol use (rates of heavy drinking, percent days abstinent), alcohol use-related self-efficacy, and intent to drink and drive. Investigators will also examine whether race/ethnicity, gender, acculturation, and alcohol situational norms predict our primary treatment outcomes (rates of heavy drinking, percent days abstinent) and DUI recidivism (alcohol-related violations).

ELIGIBILITY:
Inclusion Criteria:

* meets criteria for at-risk drinking,
* 21 years+,
* English speaking,
* current client in 3-month DUI program

Exclusion Criteria:

* under 21,
* does not speak English,
* does not meet criteria for at-risk drinking

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
heavy drinking (Survey) | 6 months
  frequency of 5 drinks per day for men and 4 drinks per day for women

SECONDARY OUTCOMES:
DUI Behaviors and Attitudes (Survey) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen C Osilla, PhD, Principal Investigator — RAND

REFERENCES:
- [Derived] Chan Osilla K, Watkins KE, Kulesza M, Florez K, Lara-Greenberg M, Miles JN. Study design to evaluate cognitive behavioral therapy among a diverse sample of adults with a first-time DUI offense. Addict Sci Clin Pract. 2016 Mar 31;11(1):7. doi: 10.1186/s13722-016-0053-x. PMID 27036221